CLINICAL TRIAL: NCT00000205
Title: Buprenorphine Maintenance Protocol
Brief Title: Buprenorphine Maintenance Protocol - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-06082-1; R18DA006082 (NIH); R18-06082-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to compare the efficacy of buprenorphine versus methadone.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Opiate dependence according to DSM-IV criteria. Self-reported use within the last 30 days. Agreeable to conditions of study and signed informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and /or nursing women. Dependence on ETOH or benzodiazepines or other sedative/hynotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1990-10; Primary Completion 1993-03 (Actual); Study Completion 1993-09 (Actual)

PRIMARY OUTCOMES:
Retention
Opiate use
Opiate craving
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Ling W, Wesson DR, Charuvastra C, Klett CJ. A controlled trial comparing buprenorphine and methadone maintenance in opioid dependence. Arch Gen Psychiatry. 1996 May;53(5):401-7. doi: 10.1001/archpsyc.1996.01830050035005. PMID 8624183
- [Background] Compton PA, Ling W, Charuvastra VC, Wesson DR. Buprenorphine as a pharmacotherapy for cocaine abuse: a review of the evidence. J Addict Dis. 1995;14(3):97-114. doi: 10.1300/J069v14n03_07. PMID 8555282
- [Background] Compton PA, Ling W, Wesson DR, Charuvastra VC, Wilkins J. Urine toxicology as an outcome measure in drug abuse clinical trials: must every sample be analyzed? J Addict Dis. 1996;15(2):85-92. doi: 10.1300/J069v15n02_07. PMID 8704003